CLINICAL TRIAL: NCT00936182
Title: A Double-Blind, Placebo-Controlled Study of the Efficacy of Fluconazole as a Treatment for Autism Spectrum Disorder
Brief Title: Study of Fluconazole in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Center for Autism and Related Disorders (Other)
Collaborators: The International Child Development Resource Center (Other); Thoughtful House (Other)
Responsible Party: Daniel Rossignol, ICDRC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0901
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fluconazole (Experimental)
  Interventions: Drug: Fluconazole
- Placebo (Placebo Comparator): Placebo capsule daily for 30 days
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Fluconazole daily for 30 days
  Other Names: Diflucan

SUMMARY:
Antifungal therapy is widely used for individuals with Autism Spectrum Disorders (ASD). The current investigation will examine the effects of fluconazole on behavioral functioning among children with ASD. This is a double-blind, randomized, placebo-controlled study of oral fluconazole in children who meet criteria for ASD. Pre- and post-treatment behavioral ratings will be used to evaluate the efficacy of fluconazole therapy. In addition, children will undergo comprehensive medical history, physical examination, and laboratory analyses.

Our objective is to quantify differences in behavioral functioning between the fluconazole treatment and a placebo. Our primary hypothesis is that, on average and relative to the placebo, children with ASD who receive fluconazole will show greater improvements in symptoms of autism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, three to ten years of age.
2. Meets clinical criteria for an autism spectrum disorder.
3. No antifungal use in the preceding 3 months.
4. Results of pyrosequencing analysis that have identified yeast
5. Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study and must provide written consent to study protocol.

Exclusion Criteria:

1. History of allergic reaction to fluconazole or other azole antifungal agents
2. Current use of terfenadine, cisapride, phenytoin, cyclosporine, rifampin, theophylline, terfenadine, cisapride, astemizole, rifabutin, or tacrolimus
3. History of uncontrolled epilepsy
4. Weight less than 15 kg at screening
5. Presence of a chronic medical condition that might interfere with study participation or where study participation would be contraindicated or clinically significant abnormal baseline laboratory results.
6. Recent (less than two months prior to study entry) initiation of behavior therapy

A child will be excluded at any point during the study if it is revealed that a major change (either addition or deletion) of treatment or service provision has occurred.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
PDD Behavior Inventory | End of study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Center for Autism and Related Disorders, Tarzana, California
  - International Child Development Resource Center, Melbourne, Florida
  - Thoughtful House, Austin, Texas